CLINICAL TRIAL: NCT03863600
Title: Validation of a Midwifery Model in Palestine
Brief Title: Midwife-led Continuity and Satisfaction With Care - an Observational Case-Control Study in Palestine
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Erik Fosse, Professor, Head of department, MD, Oslo University Hospital
Other Study IDs: Midwif 3
Record Dates: First submitted 2019-02-26; First posted 2019-03-05 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Maternal Behavior
Keywords: Satisfaction with care; Low-middle income country; Continuity of care; Maternal care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Midwife-led continuity of care: Women receiving midwife-led model of care though the continuum of pregnancy, birth and postnatal period, and who registered at the governmental clinic in a rural village.
  Interventions: Behavioral: Midwife-led continuity of care
- Regular care: Women receiving regular maternal care through the continuum of pregnancy, birth and postnatal period, and who registered at the governmental clinic in a rural village.

INTERVENTIONS:
Behavioral: Midwife-led continuity of care — Midwives from governmental hospitals provide antenatal and postnatal case-load-care in rural villages governmental clinics
  Groups: Midwife-led continuity of care

SUMMARY:
This study investigate if a midwife-led continuity model of care in Palestine, had impact on rural women's satisfaction with care through the continuum of antenatal, intrapartum and postnatal period.

DETAILED DESCRIPTION:
Between 2013 and 2016 a midwife-led continuity model of care was implemented in parts of the Palestinian governmental health system, to improve maternal services to women in rural areas on the occupied West Bank. This study investigated if and how the model influenced women's satisfaction with care, through the continuum of the antenatal-, intrapartum- and postnatal period.

Using an observational case-control design to compare the midwife-led continuity model of care with regular maternity care. Women with singleton pregnancies, who had registered for antenatal care at a rural governmental clinic, were during the first six months after birth invited to answer a questionnaire containing 60 questions with a 7-points Likert scale, rating different aspects of satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

* Residing in rural village
* Registered for pregnancy care at the villages governmental clinic
* With singleton pregnancy
* Gave birth the last one to six month

Exclusion Criteria:

* Residing in urban areas
* With multiple pregnancy
* Not registered for antenatal care at the local governmental clinic

Ages: 16 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Women who have given birth
Study Population: Rural women in the West Bank, occupied Palestine
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Mean sum-score satisfaction with care during the continuum of pregnancy,intrapartum and postnatal period | One to six months after birth
  Summarising mean score in all questions measuring satisfaction and dividing on number of questions included

SECONDARY OUTCOMES:
Mean sum-score satisfaction with care during pregnancy | One to six months after birth
  Summarising the mean score of the questions measuring satisfaction with care during pregnancy and dividing on number of questions included
Mean sum-score satisfaction with care during Labour and birth | One to six months after birth
  Summarising mean score of questions measuring satisfaction with care during Labour and birth, dividing on number of questions included
Mean sum-score satisfaction with care during postnatal period | One to six month after birth
  Summarising mean scores of questions measuring satisfaction with care during postnatal period, and dividing on number of questions included
Duration of exclusive breastfeeding | One to six month after birth
  The proportion of women who were still exclusive breastfeeding at the timepoint of interview, adjusted with number of weeks since birth

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, MD, Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Palestinian Ministry of Health, Nablus, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided
The anonymous IPD might be provided upon request

REFERENCES:
- [Derived] Mortensen B, Diep LM, Lukasse M, Lieng M, Dwekat I, Elias D, Fosse E. Women's satisfaction with midwife-led continuity of care: an observational study in Palestine. BMJ Open. 2019 Nov 3;9(11):e030324. doi: 10.1136/bmjopen-2019-030324. PMID 31685501